CLINICAL TRIAL: NCT05662943
Title: Tolerating Subretinal Fluid in Type 1 Macular Neovascularization and Polypoidal Choroidal Vasculopathy Treated Using Aflibercept
Brief Title: Outcomes of Tolerating Subretinal Fluid in Type 1 MNV and PCV
Status: Completed | Type: Observational
Sponsor: Kim's Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-09-004
Record Dates: First submitted 2022-12-09; First posted 2022-12-23 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2022-12

CONDITIONS: Polypoidal Choroidal Vasculopathy; Choroidal Neovascularization; Age-Related Macular Degeneration
Keywords: Type 1 macular neovascularization; Polypoidal Choroidal Vasculopathy; Subretinal fluid; Aflibercept; Age-related macular degeneration
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy; Choroidal Neovascularization; Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 1 Macular Neovascularization and Polypoidal Choroidal Vasculopathy: Patients with type 1 macular neovascularization and polypoidal choroidal vasculopathy who underwent continuous aflibercept injections with tolerating subfoveal retinal fluid more than 6 months
  Interventions: Drug: Intravitreal aflibercept injection

INTERVENTIONS:
Drug: Intravitreal aflibercept injection — Intravitreal injection of aflibercept (0.2 mg / 0,05 ml; Bayer Co. Ltd.,)

SUMMARY:
The purpose of the present study was to evaluate the outcomes of type 1 macular neovascularization (MNV), including polypoidal choroidal vasculopathy in patients treated tolerating subretinal fluid (SRF) using Aflibercept in a clinical setting. Approximately 150 patients are anticipated to be enrolled in this study. SRF is a primary type of fluid compartment prevalent in type 1 aneurysmal MNV. In a recent study, the prevalence of SRF during 24-month follow-up period was 36.7% to 38.8% in type 1 MNV and polypoidal choroidal vasculopathy (PCV), 20.0% in type 2 MNV, and 7.7% in type 3 MNV. In addition, patients with SRF showed better visual prognosis in type 1 MNV/PCV. For this reason, type 1 MNV is an appropriate candidate for evaluating the influence of tolerating SRF.

DETAILED DESCRIPTION:
Tolerating subretinal fluid (SRF) is one of the current major issues in the field of neovascular age-related macular degeneration. Previous post-hoc analysis studies have demonstrated that SRF is not associated with poor visual acuity as well as poor visual outcome. In addition, previous studies showed that tolerating small amount of SRF may not influence visual outcome when using treat-and-extend regimen. Based on these observations, it is generally accepted that small stable amounts of SRF can be tolerated.

To date, several clinical trials evaluated association of residual SRF with visual outcome. In these clinical trials, treatment was performed based on strict study protocol. In addition, strict rescue treatment criteria impeded definite under-treatment. However, in a clinical setting, non-scientific factors such as financial or time burden, fear to injection and compliance can influence treatment decisions. As a result, in some patients, more intensive treatment cannot be performed despite substantial amount of persistent retinal fluid.

Unlike clinical trials, in real-world practice it is difficult to precisely measure and tolerate fluid in strict amounts. As a result, large degree of fluctuation of fluid volume can occur in some patients. In addition, large amounts of fluid, which may not be tolerated in clinical trials, can persist for a relatively long period. Such cases are usually difficult to encounter in clinical trials because these patients are either treated more intensively or are dropped from the trial. Investigating the outcomes in these cases can provide useful information that cannot be obtained from clinical trials.

The purpose of the present study was to evaluate the outcomes of type 1 macular neovascularization (MNV), including polypoidal choroidal vasculopathy in patients treated tolerating SRF using Aflibercept in a clinical setting. Approximately 150 patients are anticipated to be enrolled in this study. SRF is a primary type of fluid compartment prevalent in type 1 aneurysmal MNV. In a recent study, the prevalence of SRF during 24-month follow-up period was 36.7% to 38.8% in type 1 MNV and PCV, 20.0% in type 2 MNV, and 7.7% in type 3 MNV. In addition, patients with SRF showed better visual prognosis in type 1 MNV/PCV. For this reason, type 1 MNV is an appropriate candidate for evaluating the influence of tolerating SRF.

This study may contribute to the better understanding the influence of tolerating SRF on treatment outcomes in patients diagnosed with this subtype of neovascular age-related macular degeneration (AMD). In addition, it may also contribute to the evolution of aflibercept T&E therapy, and provide evidence for physicians to guide treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Patient who were diagnosed with type 1 MNV or PCV
* Patients who were treated using aflibercept between January 2021 and December 2022
* Patients underwent continuous aflibercept injections with tolerating subfoveal retinal fluid more than 6 months.

Exclusion Criteria:

* Less than 6 months of tolerating-fluid phase
* Patients without indocyanine green angiography (ICGA) result
* Patients who received other treatment for neovascular age-related macular degeneration (AMD), except for aflibercept (eg. ranibizumab, bevacizumab, or PDT)
* History of intraocular or periocular steroid injection
* History of vitreoretinal surgery or glaucoma surgery
* History of intraocular inflammation
* Uncontrolled glaucoma (IOP ≥ 25mmHg)

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients were diagnosed with type 3 MNV or PCV and underwent continuous aflibercept injections with tolerating subfoveal retinal fluid more than 6 months
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in visual acuity | Through study completion, an average of 20 months
  Change in best-corrected visual acuity (BCVA) between the start and the end of treatment tolerating subretinal fluid

SECONDARY OUTCOMES:
Proportion of patients who exhibited deterioration of ≥0.3 logMAR BCVA | Through study completion, an average of 20 months
  Proportion of patients who exhibited deterioration of ≥0.3 logMAR BCVA between the start and the end of treatment tolerating subretinal fluid
Difference in the BCVA change, according to MNV subtype | Through study completion, an average of 20 months
  Difference in the BCVA change, according to MNV subtype (type 1 MNV vs PCV)
Degree of visual deterioration according to the treatment period | Through study completion, an average of 20 months
  Degree of visual deterioration according to the treatment period
Degree of visual deterioration according to the height of SRF | Through study completion, an average of 20 months
  Degree of visual deterioration according to the height of SRF
Degree of visual deterioration according to the fluctuation of SRF height | Through study completion, an average of 20 months
  Degree of visual deterioration according to the fluctuation of SRF height
Comparison of visual outcomes between the following three groups (mean SRF height <100 µm vs ≥100 µm, <200 µm vs ≥200 µm) | Through study completion, an average of 20 months
  Comparison of visual outcomes between the following three groups (mean SRF height <100 µm vs ≥100 µm, <200 µm vs ≥200 µm)
Risk factor of developing deterioration of ≥0.2 logMAR BCVA | Through study completion, an average of 20 months
  Risk factor of developing deterioration of ≥0.2 logMAR BCVA
Proportion of patients in whom the intraretinal fluid (IRF) developed during treatment tolerating SRF | Through study completion, an average of 20 months
  Proportion of patients in whom the IRF developed during treatment tolerating SRF
Difference in visual outcome between patients with and without IRF development | Through study completion, an average of 20 months
  Difference in visual outcome between patients with and without IRF development
Risk factors of IRF development | Through study completion, an average of 20 months
  Risk factors of IRF development
The incidence of vision-threatening event such as large submacular hemorrhage or tear of retinal pigment epithelium | Through study completion, an average of 20 months
  The incidence of vision-threatening event such as large submacular hemorrhage or tear of retinal pigment epithelium
The incidence of SRF resolution without shortening injection interval | Through study completion, an average of 20 months
  The incidence of SRF resolution without shortening injection interval

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hui Kim, M.D., Principal Investigator — Kim's Eye Hospital
Locations (1):
- Jae Hui Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sharma A, Parachuri N, Kumar N, Bandello F, Kuppermann BD, Loewenstein A, Regillo CD, Chakravarthy U. Notion of tolerating subretinal fluid in neovascular AMD: understanding the fine print before the injection pause. Br J Ophthalmol. 2021 Feb;105(2):149-150. doi: 10.1136/bjophthalmol-2020-317933. Epub 2020 Sep 26. No abstract available. PMID 32980815
- [Result] Chaudhary V, Matonti F, Zarranz-Ventura J, Stewart MW. IMPACT OF FLUID COMPARTMENTS ON FUNCTIONAL OUTCOMES FOR PATIENTS WITH NEOVASCULAR AGE-RELATED MACULAR DEGENERATION: A Systematic Literature Review. Retina. 2022 Apr 1;42(4):589-606. doi: 10.1097/IAE.0000000000003283. PMID 34393212
- [Result] Mitchell P, Holz FG, Hykin P, Midena E, Souied E, Allmeier H, Lambrou G, Schmelter T, Wolf S; ARIES study investigators. EFFICACY AND SAFETY OF INTRAVITREAL AFLIBERCEPT USING A TREAT-AND-EXTEND REGIMEN FOR NEOVASCULAR AGE-RELATED MACULAR DEGENERATION: The ARIES Study: A Randomized Clinical Trial. Retina. 2021 Sep 1;41(9):1911-1920. doi: 10.1097/IAE.0000000000003128. PMID 33782365
- [Result] Chaikitmongkol V, Sagong M, Lai TYY, Tan GSW, Ngah NF, Ohji M, Mitchell P, Yang CH, Ruamviboonsuk P, Wong I, Sakamoto T, Rajendran A, Chen Y, Lam DSC, Lai CC, Wong TY, Cheung CMG, Chang A, Koh A. Treat-and-Extend Regimens for the Management of Neovascular Age-related Macular Degeneration and Polypoidal Choroidal Vasculopathy: Consensus and Recommendations From the Asia-Pacific Vitreo-retina Society. Asia Pac J Ophthalmol (Phila). 2021 Nov 24;10(6):507-518. doi: 10.1097/APO.0000000000000445. PMID 34839342
- [Result] Cheng CK, Chen SJ, Chen JT, Chen LJ, Chen SN, Chen WL, Hsu SM, Lai CH, Sheu SJ, Wu PC, Wu WC, Wu WC, Yang CM, Yeung L, Chen TC, Yang CH. Optimal approaches and criteria to treat-and-extend regimen implementation for Neovascular age-related macular degeneration: experts consensus in Taiwan. BMC Ophthalmol. 2022 Jan 15;22(1):25. doi: 10.1186/s12886-021-02231-8. PMID 35033037
- [Result] Kim JH, Kim JW, Kim CG. Difference Between the Incidence of Retinal Fluid Subtypes and Their Association with Visual Outcomes According to the Types of Macular Neovascularization in a Korean Population. J Ocul Pharmacol Ther. 2022 Apr;38(3):261-268. doi: 10.1089/jop.2021.0103. Epub 2022 Feb 3. PMID 35119292
- [Derived] Lee JH, Kim JH. Impact of Prolonged Persisting Subretinal Fluid on the Outcome of Aflibercept Treatment in Neovascular Age-Related Macular Degeneration. J Ocul Pharmacol Ther. 2024 Mar;40(2):136-143. doi: 10.1089/jop.2023.0124. Epub 2024 Jan 12. PMID 38489060